CLINICAL TRIAL: NCT05961085
Title: Positioning of Continuous Adductor Canal Catheters After Total Knee Arthroplasty
Brief Title: Incidence of Adductor Canal Catheter Dislodgment
Status: Active, not recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 5845
Record Dates: First submitted 2023-07-11; First posted 2023-07-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adductor Canal Catheter: Pre-operative adductor canal catheter placement
  Interventions: Procedure: Adductor Canal Catheter

INTERVENTIONS:
Procedure: Adductor Canal Catheter — Ultrasound guided Adductor Canal Catheter for total knee arthroplasty analgesia

SUMMARY:
The goal of this observational study is to determine the incidence of dislodgement for adductor canal catheters after total knee arthroplasty on post-operative day 1. We will also attempt to identify factors associated with secondary catheter failure.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a common procedure for indications including osteoarthritis and malignancy involving the knee, with over 55,285 knee replacements performed between 2020-2021 in Canada. Ultrasound guided continuous adductor canal block (cACB) is the standard of care for postoperative analgesia for this procedure. The catheter is not always as effective at providing analgesia as would be expected - which could be due to displacement of the catheter. This displacement is most likely to occur peri-operatively or during physiotherapy post-operatively and as such, post-operative assessments can provide useful insight into causes of secondary failure. This prospective observational study aims to estimate the cACB dislodgment on POD 1 rate at a high volume, tertiary care referral centre, and identify factors associated with dislodgement and clinical sequelae. As this is an observational/QI study of the current standard of care at Sunnybrook Health Sciences Centre, anesthesiologists are free to use the cross sectional versus parallel insertion of the cACB per their discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for Total Knee Arthroplasty
* Older than 50 years

Exclusion Criteria:

* Body Mass Index greater than 40
* Chronic opioid consumption (greater than 30mg oral morphine equivalent daily)
* Contraindication to Adductor Canal Catheter

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to Sunnybrook Health Sciences Centre scheduled for primary total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adductor Canal Catheter tip in correct position on postoperative day 1 | Postoperative day 1 (08:00AM)
  Ultrasound confirmation of injectate spread adjacent to the femoral artery on postoperative day 1 (08h00)

SECONDARY OUTCOMES:
Adductor Canal Catheter tip in correct position after insertion | Preoperative
  Ultrasound confirmation of injectate spread adjacent to the femoral artery before surgery
Sensory block | Postoperative day 1 (08:00AM)
  Loss of sensation in the saphenous nerve distribution on postoperative day 1 (08h00)
Postoperative opioid consumption (08h00) | Postoperative day 1 (08:00AM)
  Cumulative opioid consumption after total knee arthroplasty to postoperative day 1 (08h00)
Numeric Rating Scale for Pain (NRS) at rest on postoperative day 1 (08h00) | Postoperative day 1 (08:00AM)
  Maximum pain score on 0-10 Likert Scale

OTHER OUTCOMES:
Adductor catheter occlusion | Postoperative day 1 (08:00AM)
  Any recording of local anesthetic infusion pump recording an occlusion
Patient satisfaction with analgesia on postoperative day 1 | Postoperative day 1 (08:00AM)
  Patient satisfaction measured by 0-10 Likert Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication, no limit on time
Access Criteria: Contact study investigators